CLINICAL TRIAL: NCT02306096
Title: SCAN-B: The Sweden Cancerome Analysis Network - Breast Initiative
Brief Title: Sweden Cancerome Analysis Network - Breast : Genomic Profiling of Breast Cancer
Acronym: SCAN-B
Status: Recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: South Sweden Breast Cancer Group (Unknown); Mrs. Berta Kamprad Foundation (Unknown); U-CAN (Unknown)
Responsible Party: Principal Investigator, Åke Borg, Professor, Lund University
Other Study IDs: SCANB001
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Breast Neoplasms
Keywords: prognostic and predictive biomarkers; RNA-sequencing; pathological complete response; minimal residual disease; molecular subtype; gene expression profiling; mutation screening; BRCA; translational research; genomics; transcriptomics; proteomics; metabolomics; liquid biopsy; circulating tumor cells; circulating tumor DNA; RNA-seq
MeSH Terms: conditions — Breast Neoplasms; Neoplasm, Residual; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, whole blood, serum, plasma. Collected at diagnosis and during follow-up.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the genomic profiles of breast cancer in a prospective and population-based manner. In the first phase, breast tumors are analyzed by whole transcriptome RNA-sequencing. Gene expression profiles, mutational profiles, and transcript isoform-level data will be analyzed in the context of patient information, clinicopathological variables, and outcome, with the purpose to develop new molecular diagnostic assays for breast cancer. Additional genome-scale RNA, DNA, and protein analyses will be performed in the future.

DETAILED DESCRIPTION:
Breast cancer exhibits significant molecular, pathological, and clinical heterogeneity. Current patient and clinicopathological evaluation is imperfect for predicting outcome, which results in overtreatment for many patients, and for others, leads to death from recurrent disease. Therefore, additional criteria are needed to better personalize care and maximize treatment effectiveness and survival.

The Sweden Cancerome Analysis Network - Breast (SCAN-B) study was initiated in 2010 as a multicenter prospective population-based observational study with long-sighted aims to analyze breast cancers with next-generation genomic technologies for translational research and integrated with healthcare; decipher fundamental tumor biology from these analyses; utilize genomic data to develop and validate new clinically-actionable biomarker assays; and establish real-time clinical implementation of molecular diagnostic, prognostic, and predictive tests. In the first phase, we focus on molecular profiling by next-generation RNA-sequencing. Gene expression profiles, mutational profiles, and transcript isoform-level data will be analyzed in the context of patient information, clinicopathological variables, and outcome, with the purpose to develop new molecular diagnostic assays for breast cancer. Additional genome-scale RNA, DNA, and protein analyses will be performed in the future.

As of February 2024, over 20,000 patients have enrolled in the study, representing approximately 85% of all eligible patients within the catchment region. Tissue and blood collection is integrated within healthcare routines and clinical information is provided from national quality registries.

As of Q4 2021, the SCAN-B RNA-seq analysis for molecular subtyping and risk-of-recurrence has been clinically implemented for all breast cancer patients in Skåne within the Center for Molecular Diagnostics, Laboratory Medicine, Medical Service, Region Skåne.

ELIGIBILITY:
Inclusion Criteria:

* suspicion or confirmed diagnosis of primary breast cancer
* signed informed consent

Exclusion Criteria:

* lack of signed informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suspected or confirmed diagnosis of primary breast cancer within participating hospital systems in the South Sweden Healthcare Region, Uppsala County, and Jönköping Country, Sweden. Additional hospital sites from within the Nordic countries are welcome to join.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2010-08; Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Biomarkers and clinicopathological information | up to 20-years
  Analysis of genomic data (biomarkers) and their relationship to patient and tumor clinicopathological information; assessment of analytical validity.
Invasive disease-free survival | up to 20-years
  Different biomarkers will be analysed in the context of invasive disease-free survival (IDFS) at different time-points for different subgroups of the prospective cohort, for example for all patients receiving a particular therapy or patients with tumors of a specific molecular subtype.

SECONDARY OUTCOMES:
Overall survival | 3-years, 5-years, 10-years, 15-years, 20-years
  Different biomarkers will be analysed in the context of overall survival (OS) at different time-points for different subgroups of the prospective cohort, for example for all patients receiving a particular therapy or patients with tumors of a specific molecular subtype.
Breast cancer-specific survival | 3-years, 5-years, 10-years, 15-years, 20-years
  Different biomarkers will be analysed in the context of breast cancer survival (BCS) at different time-points for different subgroups of the prospective cohort, for example for all patients receiving a particular therapy or patients with tumors of a specific molecular subtype.
Pathological response | intraoperative
  Different biomarkers will be analysed in the context of pathological response at time of surgery for patients receiving pre-operative therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Åke Borg, PhD, Study Director — Lund University; Cecilia Hegardt, PhD, Study Chair — Lund University; Christer Larsson, PhD, Principal Investigator — Lund University; Niklas Loman, MD, PhD, Principal Investigator — Skane University Hospital; Johan Vallon-Christersson, PhD, Principal Investigator — Lund University; Anna Ehinger, MD, PhD, Principal Investigator — Skane University Hospital; Lisa Rydén, MD, PhD, Principal Investigator — Skane University Hospital; Lao H Saal, MD, PhD, Principal Investigator — Lund University
Locations (9):
- Sweden (9):
  - Hallands Hospital Halmstad, Halmstad
  - Helsingborg Hospital, Helsingborg
  - Kirurgiska kliniken, Jönköping
  - Blekinge County Hospital, Karlskrona
  - Central Hospital Kristianstad, Kristianstad
  - Skåne University Hospital, Lund
  - Skåne University Hospital, Malmo
  - Uppsala University Hospital, Uppsala
  - Central Hospital Växjö, Vaxjo

IPD SHARING:
Plan to Share IPD: Undecided
Upon publication, the relevant anonymized individual participant data will be shared.

REFERENCES:
- [Background] Ryden L, Loman N, Larsson C, Hegardt C, Vallon-Christersson J, Malmberg M, Lindman H, Ehinger A, Saal LH, Borg A. Minimizing inequality in access to precision medicine in breast cancer by real-time population-based molecular analysis in the SCAN-B initiative. Br J Surg. 2018 Jan;105(2):e158-e168. doi: 10.1002/bjs.10741. PMID 29341157
- [Background] Axelsson U, Ryden L, Johnsson P, Eden P, Mansson J, Hallberg IR, Borrebaeck CAK. A multicenter study investigating the molecular fingerprint of psychological resilience in breast cancer patients: study protocol of the SCAN-B resilience study. BMC Cancer. 2018 Aug 6;18(1):789. doi: 10.1186/s12885-018-4669-y. PMID 30081937
- [Result] Saal LH, Vallon-Christersson J, Hakkinen J, Hegardt C, Grabau D, Winter C, Brueffer C, Tang MH, Reutersward C, Schulz R, Karlsson A, Ehinger A, Malina J, Manjer J, Malmberg M, Larsson C, Ryden L, Loman N, Borg A. The Sweden Cancerome Analysis Network - Breast (SCAN-B) Initiative: a large-scale multicenter infrastructure towards implementation of breast cancer genomic analyses in the clinical routine. Genome Med. 2015 Feb 2;7(1):20. doi: 10.1186/s13073-015-0131-9. eCollection 2015. PMID 25722745
- [Result] Staaf J, Glodzik D, Bosch A, Vallon-Christersson J, Reutersward C, Hakkinen J, Degasperi A, Amarante TD, Saal LH, Hegardt C, Stobart H, Ehinger A, Larsson C, Ryden L, Loman N, Malmberg M, Kvist A, Ehrencrona H, Davies HR, Borg A, Nik-Zainal S. Whole-genome sequencing of triple-negative breast cancers in a population-based clinical study. Nat Med. 2019 Oct;25(10):1526-1533. doi: 10.1038/s41591-019-0582-4. Epub 2019 Sep 30. PMID 31570822
- [Result] Vallon-Christersson J, Hakkinen J, Hegardt C, Saal LH, Larsson C, Ehinger A, Lindman H, Olofsson H, Sjoblom T, Warnberg F, Ryden L, Loman N, Malmberg M, Borg A, Staaf J. Cross comparison and prognostic assessment of breast cancer multigene signatures in a large population-based contemporary clinical series. Sci Rep. 2019 Aug 21;9(1):12184. doi: 10.1038/s41598-019-48570-x. PMID 31434940
- [Result] Dihge L, Vallon-Christersson J, Hegardt C, Saal LH, Hakkinen J, Larsson C, Ehinger A, Loman N, Malmberg M, Bendahl PO, Borg A, Staaf J, Ryden L. Prediction of Lymph Node Metastasis in Breast Cancer by Gene Expression and Clinicopathological Models: Development and Validation within a Population-Based Cohort. Clin Cancer Res. 2019 Nov 1;25(21):6368-6381. doi: 10.1158/1078-0432.CCR-19-0075. Epub 2019 Jul 24. PMID 31340938
- [Result] Lundgren C, Bendahl PO, Borg A, Ehinger A, Hegardt C, Larsson C, Loman N, Malmberg M, Olofsson H, Saal LH, Sjoblom T, Lindman H, Klintman M, Hakkinen J, Vallon-Christersson J, Ferno M, Ryden L, Ekholm M. Agreement between molecular subtyping and surrogate subtype classification: a contemporary population-based study of ER-positive/HER2-negative primary breast cancer. Breast Cancer Res Treat. 2019 Nov;178(2):459-467. doi: 10.1007/s10549-019-05378-7. Epub 2019 Aug 20. PMID 31432367
- [Result] Sokilde R, Persson H, Ehinger A, Pirona AC, Ferno M, Hegardt C, Larsson C, Loman N, Malmberg M, Ryden L, Saal L, Borg A, Vallon-Christerson J, Rovira C. Refinement of breast cancer molecular classification by miRNA expression profiles. BMC Genomics. 2019 Jun 17;20(1):503. doi: 10.1186/s12864-019-5887-7. PMID 31208318
- [Result] Persson H, Sokilde R, Hakkinen J, Pirona AC, Vallon-Christersson J, Kvist A, Mertens F, Borg A, Mitelman F, Hoglund M, Rovira C. Frequent miRNA-convergent fusion gene events in breast cancer. Nat Commun. 2017 Oct 5;8(1):788. doi: 10.1038/s41467-017-01176-1. PMID 28983113
- [Result] Persson H, Sokilde R, Hakkinen J, Vallon-Christersson J, Mitelman F, Borg A, Hoglund M, Rovira C. Analysis of fusion transcripts indicates widespread deregulation of snoRNAs and their host genes in breast cancer. Int J Cancer. 2020 Jun 15;146(12):3343-3353. doi: 10.1002/ijc.32927. Epub 2020 Feb 28. PMID 32067223
- [Result] Winter C, Nilsson MP, Olsson E, George AM, Chen Y, Kvist A, Torngren T, Vallon-Christersson J, Hegardt C, Hakkinen J, Jonsson G, Grabau D, Malmberg M, Kristoffersson U, Rehn M, Gruvberger-Saal SK, Larsson C, Borg A, Loman N, Saal LH. Targeted sequencing of BRCA1 and BRCA2 across a large unselected breast cancer cohort suggests that one-third of mutations are somatic. Ann Oncol. 2016 Aug;27(8):1532-8. doi: 10.1093/annonc/mdw209. Epub 2016 May 18. PMID 27194814
- [Result] Dahlgren M, George AM, Brueffer C, Gladchuk S, Chen Y, Vallon-Christersson J, Hegardt C, Hakkinen J, Ryden L, Malmberg M, Larsson C, Gruvberger-Saal SK, Ehinger A, Loman N, Borg A, Saal LH. Preexisting Somatic Mutations of Estrogen Receptor Alpha (ESR1) in Early-Stage Primary Breast Cancer. JNCI Cancer Spectr. 2021 Apr 22;5(2):pkab028. doi: 10.1093/jncics/pkab028. eCollection 2021 Apr. PMID 33937624
- [Result] Brueffer C, Gladchuk S, Winter C, Vallon-Christersson J, Hegardt C, Hakkinen J, George AM, Chen Y, Ehinger A, Larsson C, Loman N, Malmberg M, Ryden L, Borg A, Saal LH. The mutational landscape of the SCAN-B real-world primary breast cancer transcriptome. EMBO Mol Med. 2020 Oct 7;12(10):e12118. doi: 10.15252/emmm.202012118. Epub 2020 Sep 14. PMID 32926574
- [Result] Glodzik D, Bosch A, Hartman J, Aine M, Vallon-Christersson J, Reutersward C, Karlsson A, Mitra S, Nimeus E, Holm K, Hakkinen J, Hegardt C, Saal LH, Larsson C, Malmberg M, Ryden L, Ehinger A, Loman N, Kvist A, Ehrencrona H, Nik-Zainal S, Borg A, Staaf J. Comprehensive molecular comparison of BRCA1 hypermethylated and BRCA1 mutated triple negative breast cancers. Nat Commun. 2020 Jul 27;11(1):3747. doi: 10.1038/s41467-020-17537-2. PMID 32719340
- [Result] Larsson C, Ehinger A, Winslow S, Leandersson K, Klintman M, Dahl L, Vallon-Christersson J, Hakkinen J, Hegardt C, Manjer J, Saal L, Ryden L, Malmberg M, Borg A, Loman N. Prognostic implications of the expression levels of different immunoglobulin heavy chain-encoding RNAs in early breast cancer. NPJ Breast Cancer. 2020 Jul 6;6:28. doi: 10.1038/s41523-020-0170-2. eCollection 2020. PMID 32656317
- [Result] Fornvik D, Aaltonen KE, Chen Y, George AM, Brueffer C, Rigo R, Loman N, Saal LH, Ryden L. Detection of circulating tumor cells and circulating tumor DNA before and after mammographic breast compression in a cohort of breast cancer patients scheduled for neoadjuvant treatment. Breast Cancer Res Treat. 2019 Sep;177(2):447-455. doi: 10.1007/s10549-019-05326-5. Epub 2019 Jun 24. PMID 31236809
- [Result] Brueffer C, Vallon-Christersson J, Grabau D, Ehinger A, Hakkinen J, Hegardt C, Malina J, Chen Y, Bendahl PO, Manjer J, Malmberg M, Larsson C, Loman N, Ryden L, Borg A, Saal LH. Clinical Value of RNA Sequencing-Based Classifiers for Prediction of the Five Conventional Breast Cancer Biomarkers: A Report From the Population-Based Multicenter Sweden Cancerome Analysis Network-Breast Initiative. JCO Precis Oncol. 2018 Mar 9;2:PO.17.00135. doi: 10.1200/PO.17.00135. eCollection 2018. PMID 32913985
- [Result] Nilsson MP, Emmertz M, Kristoffersson U, Borg A, Larsson C, Rehn M, Winter C, Saal LH, Brandberg Y, Loman N. Germline mutations in BRCA1 and BRCA2 incidentally revealed in a biobank research study: experiences from re-contacting mutation carriers and relatives. J Community Genet. 2018 Jul;9(3):201-208. doi: 10.1007/s12687-017-0341-5. Epub 2017 Oct 30. PMID 29082482
- [Result] Nilsson MP, Winter C, Kristoffersson U, Rehn M, Larsson C, Saal LH, Loman N. Efficacy versus effectiveness of clinical genetic testing criteria for BRCA1 and BRCA2 hereditary mutations in incident breast cancer. Fam Cancer. 2017 Apr;16(2):187-193. doi: 10.1007/s10689-016-9953-x. PMID 28120249
- [Result] Demircan K, Bengtsson Y, Sun Q, Brange A, Vallon-Christersson J, Rijntjes E, Malmberg M, Saal LH, Ryden L, Borg A, Manjer J, Schomburg L. Serum selenium, selenoprotein P and glutathione peroxidase 3 as predictors of mortality and recurrence following breast cancer diagnosis: A multicentre cohort study. Redox Biol. 2021 Nov;47:102145. doi: 10.1016/j.redox.2021.102145. Epub 2021 Sep 21. PMID 34563873
- [Result] Dalal H, Dahlgren M, Gladchuk S, Brueffer C, Gruvberger-Saal SK, Saal LH. Clinical associations of ESR2 (estrogen receptor beta) expression across thousands of primary breast tumors. Sci Rep. 2022 Mar 18;12(1):4696. doi: 10.1038/s41598-022-08210-3. PMID 35304506
- [Result] Demircan K, Sun Q, Bengtsson Y, Seemann P, Vallon-Christersson J, Malmberg M, Saal LH, Ryden L, Minich WB, Borg A, Manjer J, Schomburg L. Autoimmunity to selenoprotein P predicts breast cancer recurrence. Redox Biol. 2022 Jul;53:102346. doi: 10.1016/j.redox.2022.102346. Epub 2022 May 25. PMID 35636018
- [Result] Staaf J, Hakkinen J, Hegardt C, Saal LH, Kimbung S, Hedenfalk I, Lien T, Sorlie T, Naume B, Russnes H, Marcone R, Ayyanan A, Brisken C, Malterling RR, Asking B, Olofsson H, Lindman H, Bendahl PO, Ehinger A, Larsson C, Loman N, Ryden L, Malmberg M, Borg A, Vallon-Christersson J. RNA sequencing-based single sample predictors of molecular subtype and risk of recurrence for clinical assessment of early-stage breast cancer. NPJ Breast Cancer. 2022 Aug 16;8(1):94. doi: 10.1038/s41523-022-00465-3. PMID 35974007
- [Result] Saghir H, Veerla S, Malmberg M, Ryden L, Ehinger A, Saal LH, Vallon-Christersson J, Borg A, Hegardt C, Larsson C, Haidar A, Hedenfalk I, Loman N, Kimbung S. How Reliable Are Gene Expression-Based and Immunohistochemical Biomarkers Assessed on a Core-Needle Biopsy? A Study of Paired Core-Needle Biopsies and Surgical Specimens in Early Breast Cancer. Cancers (Basel). 2022 Aug 18;14(16):4000. doi: 10.3390/cancers14164000. PMID 36010992
- [Result] Bengtsson Y, Demircan K, Vallon-Christersson J, Malmberg M, Saal LH, Ryden L, Borg A, Schomburg L, Sandsveden M, Manjer J. Serum copper, zinc and copper/zinc ratio in relation to survival after breast cancer diagnosis: A prospective multicenter cohort study. Redox Biol. 2023 Jul;63:102728. doi: 10.1016/j.redox.2023.102728. Epub 2023 May 16. PMID 37210781
- [Result] Demircan K, Bengtsson Y, Chillon TS, Vallon-Christersson J, Sun Q, Larsson C, Malmberg M, Saal LH, Ryden L, Borg A, Manjer J, Schomburg L. Matched analysis of circulating selenium with the breast cancer selenotranscriptome: a multicentre prospective study. J Transl Med. 2023 Sep 23;21(1):658. doi: 10.1186/s12967-023-04502-y. PMID 37741974
- [Result] Sharma A, Weitz P, Wang Y, Liu B, Vallon-Christersson J, Hartman J, Rantalainen M. Development and prognostic validation of a three-level NHG-like deep learning-based model for histological grading of breast cancer. Breast Cancer Res. 2024 Jan 29;26(1):17. doi: 10.1186/s13058-024-01770-4. PMID 38287342
- [Result] Sigurjonsdottir G, De Marchi T, Ehinger A, Hartman J, Bosch A, Staaf J, Killander F, Nimeus E. Comparison of SP142 and 22C3 PD-L1 assays in a population-based cohort of triple-negative breast cancer patients in the context of their clinically established scoring algorithms. Breast Cancer Res. 2023 Oct 10;25(1):123. doi: 10.1186/s13058-023-01724-2. PMID 37817263
- [Result] Wang Y, Ali MA, Vallon-Christersson J, Humphreys K, Hartman J, Rantalainen M. Transcriptional intra-tumour heterogeneity predicted by deep learning in routine breast histopathology slides provides independent prognostic information. Eur J Cancer. 2023 Sep;191:112953. doi: 10.1016/j.ejca.2023.112953. Epub 2023 Jun 23. PMID 37494846
- [Result] Nacer DF, Vallon-Christersson J, Nordborg N, Ehrencrona H, Kvist A, Borg A, Staaf J. Molecular characteristics of breast tumors in patients screened for germline predisposition from a population-based observational study. Genome Med. 2023 Apr 14;15(1):25. doi: 10.1186/s13073-023-01177-4. PMID 37060015
- [Result] Gulis K, Ellbrant J, Svensjo T, Skarping I, Vallon-Christersson J, Loman N, Bendahl PO, Ryden L. A prospective cohort study identifying radiologic and tumor related factors of importance for breast conserving surgery after neoadjuvant chemotherapy. Eur J Surg Oncol. 2023 Jul;49(7):1189-1195. doi: 10.1016/j.ejso.2023.03.225. Epub 2023 Mar 28. PMID 37019807
- [Result] Bjorklund SS, Aure MR, Hakkinen J, Vallon-Christersson J, Kumar S, Evensen KB, Fleischer T, Tost J; OSBREAC; Sahlberg KK, Mathelier A, Bhanot G, Ganesan S, Tekpli X, Kristensen VN. Subtype and cell type specific expression of lncRNAs provide insight into breast cancer. Commun Biol. 2022 Aug 18;5(1):834. doi: 10.1038/s42003-022-03559-7. PMID 35982125
- [Result] Sartor H, Zackrisson S, Hegardt C, Larsson C. "Association of mammographic features with molecular breast tumor profiles". Cancer Treat Res Commun. 2021;28:100387. doi: 10.1016/j.ctarc.2021.100387. Epub 2021 May 9. PMID 34004506
- [Result] Veerla S, Hohmann L, Nacer DF, Vallon-Christersson J, Staaf J. Perturbation and stability of PAM50 subtyping in population-based primary invasive breast cancer. NPJ Breast Cancer. 2023 Oct 19;9(1):83. doi: 10.1038/s41523-023-00589-0. PMID 37857634
- [Result] Aine M, Boyaci C, Hartman J, Hakkinen J, Mitra S, Campos AB, Nimeus E, Ehinger A, Vallon-Christersson J, Borg A, Staaf J. Molecular analyses of triple-negative breast cancer in the young and elderly. Breast Cancer Res. 2021 Feb 10;23(1):20. doi: 10.1186/s13058-021-01392-0. PMID 33568222
- [Derived] Mosquim Junior S, Zamore M, Vallon-Christersson J, Ryden L, Levander F. Multiomic profiling of ER-positive HER2-negative breast cancer reveals markers associated with metastatic spread. Breast Cancer Res. 2026 Jan 12. doi: 10.1186/s13058-025-02173-9. Online ahead of print. PMID 41526910
- [Derived] Sigurjonsdottir G, De Marchi T, Ehinger A, Hartman J, Ullen S, Leandersson K, Bosch A, Staaf J, Killander F, Nimeus E. Evaluation of alternative prognostic thresholds for SP142 and 22C3 immunohistochemical PD-L1 expression in triple-negative breast cancer: results from a population-based cohort. Breast Cancer Res Treat. 2025 Apr;210(2):271-284. doi: 10.1007/s10549-024-07561-x. Epub 2024 Dec 10. PMID 39656429
- [Derived] Rediti M, Venet D, Joaquin Garcia A, Maetens M, Vincent D, Majjaj S, El-Abed S, Di Cosimo S, Ueno T, Izquierdo M, Piccart M, Pusztai L, Loi S, Salgado R, Viale G, Rothe F, Sotiriou C. Identification of HER2-positive breast cancer molecular subtypes with potential clinical implications in the ALTTO clinical trial. Nat Commun. 2024 Nov 29;15(1):10402. doi: 10.1038/s41467-024-54621-3. PMID 39613746
- [Derived] Fornvik D, Borgquist S, Larsson M, Zackrisson S, Skarping I. Deep learning analysis of serial digital breast tomosynthesis images in a prospective cohort of breast cancer patients who received neoadjuvant chemotherapy. Eur J Radiol. 2024 Sep;178:111624. doi: 10.1016/j.ejrad.2024.111624. Epub 2024 Jul 14. PMID 39029241
- See also: Sweden Cancerome Analysis Network - Breast (SCAN-B) Website (Lund University) [SWEDISH LANGUAGE] — https://www.scan-b.lu.se
- Available data/document: RNA-seq Processed Gene Expression Data and Annotations (n=49 patients): GSE60789 — https://www.ncbi.nlm.nih.gov/geo/query/acc.cgi?acc=GSE60789 — SuperSeries: GSE60789 SubSeries: GSE60785, GSE60788
- Available data/document: RNA-seq Processed Gene Expression Data and Annotations (n=3678 patients): GSE81540 — https://www.ncbi.nlm.nih.gov/geo/query/acc.cgi?acc=GSE81540 — SuperSeries: GSE81540 SubSeries: GSE81538, GSE96058